CLINICAL TRIAL: NCT03470636
Title: Clinical Study of the HeartLight X3 Endoscopic Ablation System (EAS) With Excalibur Balloon Compared to HeartLight System in the Treatment of Symptomatic Atrial Fibrillation
Brief Title: Clinical Study of the HeartLight X3 Endoscopic Ablation System With Excalibur Balloon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-4378
Record Dates: First submitted 2018-03-06; First posted 2018-03-20 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HeartLight X3 (Experimental): Pulmonary vein isolation using HeartLight X3
  Interventions: Device: HeartLight X3

INTERVENTIONS:
Device: HeartLight X3 — Pulmonary vein isolation

SUMMARY:
The objective of the study is to demonstrate the improved ablation and procedure times of the HeartLight X3 compared to the current HeartLight catheter in the treatment of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal atrial fibrillation failure of at least one AAD others

Exclusion Criteria:

* overall good health as established by multiple criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Ablation time | Acute - at the end of the index procedure
  Ablation time

SECONDARY OUTCOMES:
Procedure time | Acute - at the end of the index procedure
  Procedure time
PV Isolation | Acute - at the end of the index procedure
  Percent of isolated pulmonary veins
PAE Rate | 30 Days
  Primary Adverse Event rate
AF Free Rate | 6 and 12 months
  6- and 12-month chronic results

CONTACTS AND LOCATIONS:
Overall Officials: Burke T. Barrett, Study Director — CardioFocus, Inc.
Locations (1):
- Nemocnice Na Homolce, Prague, Czechia

REFERENCES:
- [Derived] Schmidt B, Petru J, Chun KRJ, Sediva L, Bordignon S, Chen S, Neuzil P. Pivotal Study of a Novel Motor-Driven Endoscopic Ablation System. Circ Arrhythm Electrophysiol. 2021 Mar;14(3):e009544. doi: 10.1161/CIRCEP.120.009544. Epub 2021 Feb 11. PMID 33570423